CLINICAL TRIAL: NCT00691925
Title: Contact Lens for Mitigating Pain Following Refractive Procedure
Brief Title: Mitigating Pain Following Refractive Surgery
Status: Completed | Type: Observational
Sponsor: FORSIGHT Vision3 (Industry)
Responsible Party: Osnat Ehrman, FORSIGHT
Other Study IDs: 0164
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 2009-06

CONDITIONS: Pain
Keywords: refractive surgery
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: bilateral post refractive surgery subject

SUMMARY:
Using Contact lens following refractive procedure to reduce pain.

DETAILED DESCRIPTION:
Patients at day 1 following the procedure will be treated with a contact lens and assessed for pain at 1,2,4 hours and 1,3,5 days.

prospective comparative study

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent bilateral Refractive surgery for myopic correction.
2. Age 18-60.
3. Evidence of an epithelial defect.
4. Patient complains of significant pain.
5. Patients able to understand the requirements of the study and willing to follow study instructions, to provide written informed consent to participate, and who agree to comply with all study requirements, including the required study follow-up visits.

Exclusion Criteria:

1. Any other anterior segment abnormality other than that associated with Refractive surgery.
2. Any abnormalities associated with the eye lids.
3. Prior laser treatment of the retina.
4. Any ophthalmic surgery performed within three (3) months prior to study excluding Refractive surgery.
5. Diagnosis of glaucoma.
6. Active diabetic retinopathy.
7. Clinically significant inflammation or infection within six (6) months prior to study.
8. Uncontrolled systemic disease (e.g., diabetes, hypertension, etc.) in the opinion of the Investigator.
9. Participation in any study involving an investigational drug within the past 30 calendar days, or ongoing participation in a study with an investigational material.
10. Intolerance or hypersensitivity to topical anesthetics,
11. Specifically known intolerance or hypersensitivity to contact lenses.
12. A medical condition, serious intercurrent illness, or extenuating circumstance that would significantly decrease study compliance, including all prescribed follow-up.
13. Any condition that, in the opinion of the investigator, would jeopardize the safety of the patient.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: at least 10 subjects following refractive surgery
Sampling Method: Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2008-06; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Verssano, MD, Principal Investigator — Sorasky Medical Center
Locations (1):
- Sorasky Medical Center, Tel Aviv, Israel